

### ClinicalTrials.gov Protocol Registration and Results System (PRS) Receipt

Release Date: May 29, 2024

#### ClinicalTrials.gov ID: [Not yet assigned]

# Study Identification

Unique Protocol ID: IIT2023015

Brief Title: Comparison of Short-term and Long-term Outcomes of Robotic and

Laparoscopic Right Colon Cancer: a 10-year Single-center Large-sample

Retrospective Study

Official Title: the Ethics Committee of the First Affiliated Hospital of Nanchang University

Secondary IDs:

## **Study Status**

Record Verification: May 2024 Overall Status: Completed

Study Start: December 1, 2014 [Actual] Primary Completion: March 31, 2024 [Actual] Study Completion: April 30, 2024 [Actual]

## Sponsor/Collaborators

Sponsor: Taiyuan Li

Responsible Party: Sponsor-Investigator

Investigator: Taiyuan Li [tli]

Official Title: the First Affiliated Hospital of Nanchang University

Affiliation: Nanchang University

Collaborators:

# **Oversight**

U.S. FDA-regulated Drug: No U.S. FDA-regulated Device: No

U.S. FDA IND/IDE: No

Human Subjects Review: Board Status: Exempt

Data Monitoring:

## **Study Description**

Brief Summary: The goal of this observational study is to evaluate the short-term outcomes and

long-term outcomes of robot-assisted right colon group for cancer compared

to laparoscopic-assisted right colon group. This is a large sample study based on ten years of clinical data. The main question it aims to answer is: What are the advantages of da Vinci robot right hemicolectomy compared to laparoscopic right hemicolectomy, and is there a difference in long-term efficacy between the two methods.

**Detailed Description:** 

### **Conditions**

Conditions: Robotic, Laparoscopic, Colon Cancer, Short-term Outcomes, Long-term

Outcomes

Keywords:

# **Study Design**

Study Type: Observational

Observational Study Model: Cohort

Time Perspective: Retrospective

Biospecimen Retention: Biospecimen Description:

Enrollment: 1879 [Actual]

Number of Groups/Cohorts: 2

# **Groups and Interventions**

| robot-assisted right colon group | |
|---|---|
| Robot assisted radical surgery for right colon cancer | Device: Da Vinci Robot Surgical System Performing surgery on right colon cancer patients using the da Vinci robotic surgical system or laparoscopic surgical system |
| laparoscopic-assisted right colon group Laparoscopic assisted radical surgery for right colon cancer | Other Names: • Laparoscopic surgical system Device: Da Vinci Robot Surgical System Performing surgery on right colon cancer patients using the da Vinci robotic surgical system or laparoscopic surgical system Other Names: • Laparoscopic surgical system |

### **Outcome Measures**

Primary Outcome Measure:

- 1. overall survival [Time Frame: months]
- 2. disease-free survival

[Time Frame: months]

#### Secondary Outcome Measure:

3. the rate of postoperative complications

[Time Frame: rates]

4. operative time

[Time Frame: minute]

5. estimation of blood loss

[Time Frame: ml]

6. number of retrieved lymph nodes

[Time Frame: Number]

7. days after postoperative hospital stay

[Time Frame: day]

8. time to first exhaust

[Time Frame: hours]

9. time to liquid diet [Time Frame: hours]

10. the rate of intracorporeal anastomosis

[Time Frame: rates]

# **Eligibility**

Study Population: The consecutive cases of robotic-assisted or laparoscopic-assisted right

colectomy between December 2014 and March 2024. All cases derived from

the First Affiliated Hospital of Nanchang University.

Sampling Method: Non-Probability Sample

Minimum Age: 18 Years Maximum Age: 85 Years

Sex: All

Gender Based:

Accepts Healthy Volunteers: No

Criteria: Inclusion Criteria:1) age: 18-85 years; 2) no distant metastasis; 3) preoperative

colonoscopy showing that the tumor was located in the ileocecal region, ascending colon, hepatic flexure, or transverse colon with pathology showing

malignancy; 4) signed informed consent.

\_

Exclusion Criteria:1) multiple primary colorectal cancer; 2) recurrent right colon cancer; 3) preoperative neoadjuvant chemotherapy; 4) emergency surgery for intestinal obstruction, bleeding or perforation; 5) incomplete data and missing

follow-up data.

-

#### Contacts/Locations

Central Contact Person: Taiyuan Li, doctor

Email: ndyfy00530@ncu.edu.cn

Central Contact Backup: shanping Ye, doctor

| | Email: ndyfy08807@ncu.edu.cn |
|------------------|------------------------------|
| Study Officials: | |
| Locations: | |

# **IPDSharing**

Plan to Share IPD: Undecided

Access to the database can be obtained from the corresponding author on

reasonable request.

## References

Citations:

Links:

Available IPD/Information:

U.S. National Library of Medicine | U.S. National Institutes of Health | U.S. Department of Health & Human Services